CLINICAL TRIAL: NCT04394689
Title: A Phase I/II, Double-blind, Randomized, Active-controlled, Age De-escalation Trial to Assess Safety and Immunogenicity of a Measles Rubella Vaccine (MRV) Microneedle Patch (MRV-MNP) in Adults, MRV-primed Toddlers, and MRV-naïve Infants
Brief Title: Measles and Rubella Vaccine Microneedle Patch Phase 1-2 Age De-escalation Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Micron Biomedical, Inc (Industry)
Collaborators: Medical Research Council (Other Government); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SCC22420
Record Dates: First submitted 2020-05-06; First posted 2020-05-19 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Measles; Rubella; Vaccination; Healthy
Keywords: Rubella vaccine safety; Measles vaccine safety; Microneedle patch
MeSH Terms: conditions — Measles; Rubella

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of two arms: Active Comparator (subcutaneous measles rubella vaccine [MRV] via needle and syringe [SC]), or MRV as a microneedle patch [MNP].
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, care provider, and investigator blinding will occur through use of a double-dummy design; subjects randomized to the MRV-MNP group will also receive a placebo (PLA) saline injection, and subjects randomized to the MRV-SC group will also receive a PLA-MNP.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRV-SC (Active Comparator): A standard, single dose of Measles Rubella vaccine delivered subcutaneously with a needle and syringe
  Interventions: Biological: Measles Rubella Vaccine (MRV-SC); Other: PLA-MNP
- MRV-MNP (Experimental): A single dose of Measles Rubella vaccine delivered intradermally with a microneedle patch
  Interventions: Biological: MRV-MNP; Other: PLA-SC

INTERVENTIONS:
Biological: Measles Rubella Vaccine (MRV-SC) — One dose as subcutaneous injection of a WHO prequalified MR vaccine
  Arms: MRV-SC
Biological: MRV-MNP — One standard dose of Measles and Rubella vaccine delivered intradermally as a dissolving microneedle patch
  Arms: MRV-MNP
Other: PLA-MNP — One placebo dose of a dissolving microneedle patch
  Arms: MRV-SC
Other: PLA-SC — Placebo saline as subcutaneous injection
  Arms: MRV-MNP

SUMMARY:
This is a phase 1/2, single-centre, double-blind, double-dummy, randomized, active-controlled, age de-escalation trial. Age de-escalation will be based on a review of the safety data from the preceding cohort (adults for toddlers and toddlers for infants) up to day 14 post study product administration by a data monitoring committee (DMC). All participants will receive either the MRV-MNP and a placebo (0.9% sodium chloride) SC injection (PLA-SC) or a placebo-MNP (PLA-MNP) and MRV by the SC route (MRV-SC). Only those study staff randomizing participants and preparing the study products for administration will be aware of the products administered. Those administering the study products, all other trial staff and the participants and parents will be blinded to treatment group. 45 adults (18 to 40-years-of-age) will be randomized in a 2:1 ratio. Thus, 30 adults will receive MRV-MNP and PLA-SC while 15 adults will receive MRV-SC and PLA-MNP. 120 toddlers (15 to 18 months-of-age) will be randomized in a 1:1 ratio. Thus, 60 toddlers will receive MRV-MNP and PLA-SC while the same number of toddlers will receive MRV-SC and PLA-MNP. 120 infants (9 to 10 months) will also be randomized in a 1:1 ratio. Thus, 60 infants will receive MRV-MNP and PLA-SC while the same number of infants will receive MRV-SC and PLA-MNP. Solicited local and systemic AE will be collected daily from all participants from the day of study product administration to day 13 post study product administration. Unsolicited AE and SAE will be collected from the day of study product administration to day 180 post study product administration. All participants will have laboratory investigations (hepatitis B, hepatitis C, hematology and biochemistry) conducted as part of screening. Adults will have safety laboratory investigations repeated on day seven and day 14 post study product administration. Toddlers and infants will have safety laboratory investigations repeated on day seven post study product administration. All participants will have measles- and rubella-specific SNA titers and measles- and rubella-specific IgG concentrations measured at baseline and day 42 and 180 post study product administration. Other Expanded Program on Immunization (EPI) vaccines due in toddler (oral poliovirus vaccine, diphtheria-tetanus-pertussis) and in infants (oral poliovirus vaccine, yellow fever vaccine and MenAfriVac® [due at 12 months]) will be given by the investigator team at the day 42 study visit (V4).

ELIGIBILITY:
Inclusion Criteria:

* Adults: Be between 18 and 40 years inclusive on the day of consent.
* Toddlers: Be between 15 and 18 months of age inclusive on the day of consent.
* Infants: Be between 9 and 10 months of age inclusive on the day of consent.
* Be judged to be able to comprehend and comply with study requirement and procedures and must be willing and able to return for all scheduled follow-up visits (adult cohort).
* Have a parent who is judged to be able to comprehend and comply with study requirement and procedures and is willing and able to return for all scheduled follow-up visits (toddler and infant cohort).
* Be willing to avoid consumption (ingestion and topical application) of herbal or other local traditional medications throughout the course of the study.
* Have a readily identifiable place of residence within a reasonable travelling distance of the clinical trial site.
* Have a consistent means of telephone contact for the duration of trial participation
* Have a site on one wrist that is judged to be suitable for MNP administration.
* Adult female cohort only: have a negative serum pregnancy test at screening (V0) and negative urine pregnancy test on the day of vaccination (V1).
* Adult female cohort only: employ an effective method of birth control for two months preceding and throughout the study
* Toddler cohort only: have been parenterally vaccinated against measles and rubella at between nine and 12 months of age.

Exclusion Criteria:

* Have used any investigational product within the 90 days prior to study product administration or plan to use any investigational products during the period of study participation.
* Have consumed (by ingestion or topical application) any herbal or other traditional medication within 14 days of study product administration
* Have a history of serious reactions to any prior vaccination or known hypersensitivity to any component of the MRV-MNP, MRV-SC or PLA-MNP including polyethylene foam with acrylic adhesive, silicone-coated Kraft paper, stainless steel, and severe allergic reactions to cow's milk.
* Have a history of anaphylactic shock or other life-threatening allergic reactions
* Have any chronic, clinically significant pulmonary, cardiovascular, hepatobiliary, gastrointestinal, renal, neurological, or haematological abnormality or illness that requires medical therapy.
* Have a history of administration of any non-study vaccines within the 56 days before the administration of study products or planned vaccination during study participation, except for non-measles and rubella catch-up/national campaign administered through the Gambian Ministry of Health.
* Have a history of chronic administration (defined as more than 14 consecutive days) of immunosuppressant (> 0.5mg/kg/day of prednisolone or equivalent) or other immune modifying drugs within the 12 months prior to the administration of the study vaccine including the use of glucocorticoids. The use of inhaled/per nasal glucocorticoids will be permitted. The use of topical glucocorticoids within 12 months is not permitted.
* Have a history of the administration of immunoglobulins and/or any blood products within the 12 months prior to administration of the study vaccine or anticipation of such administration during the study period.
* Have a history of known disturbance of coagulation or blood disorder that could cause anaemia or excess bleeding (e.g. sickle cell disorders, thalassemia, and coagulation factor deficiencies).
* Have a history of keloid formation.
* Have significant scars, tattoos, rashes or other dermatologic condition in the area of the vaccination site which will interfere with the application of the MNP and assessment of local solicited AE.
* Have human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection based on screening laboratory investigations.
* Have any medical or social condition that in the opinion of the study clinician may interfere with the study objectives, pose a risk to the participant, or prevent the participant from completing the study follow-up.
* Be an employee of, or direct descendant (child or grandchild) of any person employed by the investigator or sponsor.
* Have plans to travel outside the study area for an extended duration during the period of study participation.
* Have any screening laboratory test with a toxicity score of ≥ 2 or with a toxicity score of 1 which is nonetheless judged to be clinically significant by the trial clinician.
* Have any vital sign (heart rate, respiratory rate, non-invasive blood pressure [adult cohort only]) with a toxicity score of > 1.
* Have an axillary temperature of > 37.5°C and have had a documented fever at the same level in the 72 hours preceding randomization and vaccination.
* Have a history of an illness with a fever and rash suggestive of measles in the preceding two months.
* Have any acute illness (severity grade > 2).
* Have a positive rapid diagnostic test (RDT) (or blood film) for malaria.
* Adult cohort only: Have been vaccinated against measles or rubella in the preceding four years.
* Adult cohort only: Have a BMI of < 18.5kg/m2 (underweight) or > 35kg/m2 (severely obese).
* Adults cohort only: Have a recent history (within the past year) or signs of alcohol or substance abuse.
* Adult cohort only: Have a history of major psychiatric disorder.
* Adult cohort only: Have a history of blood donation within three months of study enrollment or plans to donate blood during participation in the study.
* Adult female cohort only: Be pregnant or breast-feeding.
* Toddler and infant cohort only: Have been vertically exposed to HIV based on maternal history.
* Toddler and infant cohorts only: Have a weight for height z-score below -2SD (moderate malnutrition).
* Infant cohort only: Have been vaccinated against measles or rubella.

Ages: 9 Months to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 281 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent solicited adverse events as assessed by the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (V2.1 Jul 2017) | 14 days
  The number, severity and relatedness of solicited local and systemic adverse events collected on the day of study product administration and daily until day 14 following study product administration.
Incidence of pan-study unsolicited adverse events, as assessed by the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events. | 180 days
  The number, severity and relatedness of unsolicited adverse events and serious adverse events from the day of study product administration until day 180 following study product administration.
Incidence of treatment-emergent biochemical and hematological abnormalities as assessed by regional laboratory normal values for a given test | up to 14 days
  The number, severity and relatedness of biochemical and hematological abnormalities occurring until day 14 (Adult cohort only), or day 7 (toddler and infant cohorts) following study product administration.

SECONDARY OUTCOMES:
Percentage of measles seroprotected participants | Days 42 and 180 post vaccination
  Measles serum neutralization antibody (SNA) titers by plaque reduction neutralization test (PRNT). Measles serum IgG binding antibody concentrations by a bead-based multiplex assay. Measles seropositivity will be defined as a standardized titer of ≥ 200mIU/mL.
Percentage of rubella seroprotected participants | Days 42 and 180 post vaccination
  Rubella SNA titers by indirect immunocolorimetric assay (ICA). Rubella serum IgG binding antibody concentrations by a bead-based multiplex assay. Rubella seropositivity will be defined as a standardized titer of ≥ 10IU/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Ed Clarke, MD, Principal Investigator — Medical Research Center, The Gambia
Locations (1):
- Medical Research Center The Gambia at LSHTM, Fajara, The Gambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adigweme I, Akpalu E, Yisa M, Donkor S, Jarju LB, Danso B, Mendy A, Jeffries D, Njie A, Bruce A, Royals M, Goodson JL, Prausnitz MR, McAllister D, Rota PA, Henry S, Clarke E. Study protocol for a phase 1/2, single-centre, double-blind, double-dummy, randomized, active-controlled, age de-escalation trial to assess the safety, tolerability and immunogenicity of a measles and rubella vaccine delivered by a microneedle patch in healthy adults (18 to 40 years), measles and rubella vaccine-primed toddlers (15 to 18 months) and measles and rubella vaccine-naive infants (9 to 10 months) in The Gambia [Measles and Rubella Vaccine Microneedle Patch Phase 1/2 Age De-escalation Trial]. Trials. 2022 Sep 14;23(1):775. doi: 10.1186/s13063-022-06493-5. PMID 36104719